CLINICAL TRIAL: NCT05986721
Title: A Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of AGB101 on Slowing Progression of Mild Cognitive Impairment Due to Alzheimer's Disease in Apolipoprotein E4 Non-carriers
Brief Title: Clinical Trial of AGB101 for Mild Cognitive Impairment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: AgeneBio (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGB101 NE4
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment; Prodromal Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Levetiracetam

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 2:1, 3:1, or 4:1, following an escalating randomization scheme. A total of 60 subjects will be randomized (approximately 44 subjects will be randomized to AGB101 and 16 to placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Oral Tablet (Placebo Comparator): Matching placebo to AGB101 tablet once daily, taken orally, for 78 weeks
  Interventions: Drug: Placebo
- AGB101 220 mg tablet (Experimental): Single 220 mg AGB101 tablet once daily, taken orally, for 78 weeks.
  Interventions: Drug: AGB101

INTERVENTIONS:
Drug: AGB101 — low-dose levetiracetam, 220 mg, extended release tablet
  Other Names: levetiracetam; keppra
  Arms: AGB101 220 mg tablet
Drug: Placebo — Placebo oral tablet
  Other Names: placebo tablet
  Arms: Placebo Oral Tablet

SUMMARY:
The primary objective of the study is to evaluate the efficacy of AGB101 on slowing cognitive and functional impairment as measured by reduction in neuronal injury in participants with mild cognitive impairment due to Alzheimer's Disease. Participants will be randomized to receive placebo or AGB101 (220 mg), once daily for 78 weeks. Secondary objectives are to assess the effect of AGB101 compared with placebo on clinical progression as measured by the Clinical Dementia Rating Scale- Sum of Boxes and Memory Box score.

DETAILED DESCRIPTION:
AGB101 is hypothesized to slow the progression of MCI due to AD by restoring the entorhinal/hippocampal network balance. During this phase of the disease, fMRI studies show hippocampal over-activity and EC under-activity. As shown in the phase 2 study, AGB101 restores this network balance by attenuating hippocampal over-activity and restoring EC activity. Hippocampal over-activity predicts progression on EC atrophy (primary endpoint) and on CDR-SB (secondary endpoint). By restoring network balance, AGB101 is hypothesized to improve cognitive function (CDR-SB) and reduce neuronal injury (EC atrophy).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 55 and 85 years old (inclusive) in good general health:

   1. Willing and able to consent and participate for the duration of the study.
   2. Have eighth-grade education or good work history sufficient to exclude mental retardation.
   3. Have visual and auditory acuity adequate for neuropsychological testing.
   4. Have proficient fluency of the native local language to participate in all the neuropsychological test assessments.
2. Have a study partner who has sufficient contact with the subject to be able to provide assessment of memory changes, who can accompany the subject to the screening visit and all major clinic visits for the duration of those visits, and who is able to provide an independent evaluation of the subject's functioning.
3. Have MCI as defined by all of the following criteria and consistent with the National Institute on Aging-Alzheimer's Association criteria:

   1. MMSE scores between 24 and 30 (inclusive; exceptions may be made for subjects with <8 years of education at the discretion of the sponsor).
   2. A memory complaint reported by the subject or his/her study partner.
   3. Evidence of lower memory performance based on the delayed recall portion on a list learning task (ISLT or BSRT).
   4. A CDR score of 0.5 with a memory box score of ≥ 0.5.
   5. Essentially preserved activities of daily living.
   6. Cognitive decline not primarily caused by vascular, traumatic, or medical problems (alternative causes of cognitive decline are ruled out).
4. Have an Apolipoprotein E (ApoE) genotype that does not include one or more E4 alleles.
5. Permitted medications:

   1. With potential pro-cognitive effects, such as cholinesterase inhibitors and memantine, must be at a stable dose for ≥ 3 months prior to screening and expected to remain stable throughout the study; estrogen replacement therapy, Ginkgo biloba, and vitamin E must be at a stable dose for ≥ 4 weeks prior to screening and expected to remain stable throughout the study.
   2. Other psychotropics, such as antidepressants and antipsychotics, must be at a stable dose for ≥ 3 months prior to screening and expected to remain stable throughout the study.
6. Willing and able to undergo imaging procedures:

   1. An amyloid-imaging PET scan with 11C-PiB or documented evidence of an amyloid-positive PET scan.

      The amyloid PET scan performed at baseline must be read by a qualified physician with experience in reading amyloid PET scans, and it should be consistent with the presence of amyloid plaques.
   2. Repeated MRI scans (3 Tesla) with no contraindications to MRI. The MRI scan performed at baseline must be read by a physician with experience in evaluating brain-imaging studies in dementia. MRI scan results are consistent with the diagnosis of amnestic MCI due to AD with no clinically significant findings of non-AD pathology that could account for the observed cognitive impairment.
7. Willing to allow collection of blood for apolipoprotein E (ApoE) genotyping and banking.

Exclusion Criteria:

1. Carrying one or more copies of the apolipoprotein E4 (ApoeE4) allele.
2. Use of anticonvulsant medications or excluded psychotropic medications within 3 months prior to the baseline visit.
3. Use of anti-amyloid medications at any time prior to screening visit, or at any time during the study.
4. Participation in a therapeutic clinical study for any medical or psychiatric indications within 3 months (6 months for biologics) of the screening visit, or at any time during the study. Subjects must understand that they may only enroll in this clinical study once; they may not enroll in any other clinical study while participating in the current study, and they may not participate in a clinical study of a drug, biologic, therapeutic device, or medical food, in which the last dose/administration was received within 3 months (6 months for biologics) prior to screening.
5. History of hypersensitivity or lack of tolerability to AGB101 (levetiracetam).
6. Severe renal impairment (creatinine clearance of < 30 mL/minute) or undergoing hemodialysis.
7. Any significant neurological disease other than suspected incipient AD, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder (lifetime history; infant febrile seizures are not exclusionary), subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits, or known structural brain abnormalities.
8. Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, or body that constitute a contraindication to having an MRI.
9. Diagnosis of bipolar disorder, or major depression within the past 3 years, as described in the DSM-5. Psychotic features, agitation, or behavioral problems within the last 3 months that could lead to difficulty complying with the protocol. Subjects must not have a major depressive disorder or other types of depression that could confound diagnosis of MCI due to AD, or clinical assessments, in the opinion of the investigator. The Geriatric Depression Scale [GDS] (long form score > 9 suggests depression) results should be reviewed by the investigator to assist in this determination.
10. Modified Hachinski Ischemic Scale (HIS) score > 4.
11. History of schizophrenia (DSM-5 criteria).
12. History of alcohol or substance abuse or dependence within the past 3 years (DSM-5 criteria).
13. Any significant systemic illness or unstable medical condition that could lead to difficulty in complying with the protocol requirements.
14. Any unstable medical condition that is likely to require new medical or surgical treatment during the course of the study and where such treatments might affect the collection of efficacy data.
15. Clinically significant abnormalities in B12 or thyroid function test that might interfere with the study. A low B12 (below normative range for elderly) is exclusionary, unless follow-up labs (homocysteine and methylmalonic acid) indicate that it is not physiologically significant. If the B12 deficiency is treated, subjects may become eligible to participate in the study.
16. Residence in a skilled nursing facility. Individuals in independent living communities, assisted living facilities, residential care facilities, or continuing care communities are eligible provided they engage in a sufficient spectrum of activity to permit assessment of all 6 domains contributing to the CDR-SB. Individuals in these facilities must also have a study partner who has the ability to observe the subject during the study and can participate in clinical evaluations.
17. Any use of excluded medications (eg, antiepileptics, certain antidepressants or antipsychotics, antihistamines with anticholinergic properties, opiates).
18. Participation in clinical studies using the ISLT/BSRT, BPS-O task, or the trail making test (A, B) within 1 month of screening.
19. Female subjects must not be pregnant, lactating, or of childbearing potential (ie, they must be 2 years postmenopause or surgically sterile).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Entorhinal Cortex (EC) Volume From Baseline | 78 weeks
  Magnetic resonance imaging (MRI) will be used to assess neuronal injury via change in EC volume from baseline to 78 weeks. Negative change scores indicate reduced volume at 78 weeks and positive change scores indicate increase in volume at 78 weeks. Greater numbers therefore correspond with better outcomes.

SECONDARY OUTCOMES:
Change in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) Score From Baseline | 78 weeks
  CDR-SB scores at baseline will be subtracted from CDR-SB scores at week 78 to generate the change score from baseline, with a possible total range of -18 to 18. Positive change scores reflect greater impairment on the CDR-SB at week 78, while negative change scores reflect less impairment on the CDR-SB at week 78.
Change in Clinical Dementia Rating Scale - Memory Box Score From Baseline | 78 weeks
  The CDR- memory box score at baseline will be subtracted from the CDR- memory box score at week 78 to generate the change score from baseline, with a possible total range of -3 to 3. Positive change scores reflect greater impairment on the CDR-SB at week 78, while negative change scores reflect less impairment on the CDR-SB at week 78.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No